CLINICAL TRIAL: NCT02809040
Title: E_Stethoscope : Portable Digital Auscultation Based on Wireless Sensor Node to Diagnose Diastolic Dysfunction in Hypertensive Heart Disease
Brief Title: E_Stethoscope: Portable Digital Auscultation Study on Hypertensive/Hypertensive Heart Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/2083
Record Dates: First submitted 2016-05-31; First posted 2016-06-22 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Hypertension; Hypertensive Heart Disease
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hypertensive Heart Disease: Portable Digital Auscultation/ Electrocardiogram/Echocardiography/ Traditional Stethoscope
  Interventions: Other: Electrocardiogram/Echocardiography; Other: Portable digital auscultation
- Volunteer subjects: Portable Digital Auscultation/ Electrocardiogram/Echocardiography/ Traditional Stethoscope
  Interventions: Other: Electrocardiogram/Echocardiography; Other: Portable digital auscultation
- Diagnosed Hypertension: Portable Digital Auscultation/ Electrocardiogram/Echocardiography/ Traditional Stethoscope
  Interventions: Other: Electrocardiogram/Echocardiography; Other: Portable digital auscultation

INTERVENTIONS:
Other: Electrocardiogram/Echocardiography — Electrocardiogram (ECG) is a non-invasive (does not require an incision into the body) test that records the electrical activity of the heart.
  Echocardiography is a non-invasive scanning of heart images using standard two-dimensional, three-dimensional, and Doppler ultrasound to create images of the heart.
Other: Portable digital auscultation — Traditional Stethoscope :An acoustic medical device for auscultation, or listening to internal sounds of human body.
  Digital Stethoscope :Electronic stethoscope is a passive heart sound recording device. The heart sound listening and recording will be performed by trained personnel in a way very similar to that of using conventional cardiac auscultation

SUMMARY:
Hypertensive heart disease (HHD) is a heart condition that is caused by chronic exposure to high blood pressure. In patients with HHD, abnormalities in the way heart muscle relaxes and how heart chambers passively fill with blood (diastolic dysfunction) can occur that may be detected on echocardiography (echo), which is a standard clinical method to examine heart structure and function using reflected sound waves. Investigators propose to develop a digital auscultation system or electronic stethoscope based on wireless sensor node technique. Investigators hypothesize that the heart sounds measurements detected by electronic stethoscope can be used to detect heart diastolic dysfunction in HHD .

DETAILED DESCRIPTION:
Study proposal aims to look into treatment of hypertension (HT) and its complications of the exact high healthcare costs. In 2004, Singapore adult prevalence of hypertension was 20.1%. World Health Organization estimates that HT causes 4.5% of global disease burden, and that 62% of cerebrovascular disease and 49% of ischemic heart disease are attributable to suboptimal blood pressure (BP) control.

Recently, scrutiny has been focused on appropriate BP levels at which to initiate HT treatment with the benefit of strict BP targets in otherwise uncomplicated HT is questioned, as HT drug treatment is not without risks. This underscores the need to stratify hypertension patients according to target organ damage, so that affected HT patients may be selected for intensive BP lowering.

Hypertensive heart disease (HHD) is a heart condition that is caused by chronic exposure to high BP. As population ages, both HT and Hypertensive Heart Disease prevalence increase. Genetic and hemodynamic factors interact to cause Hypertensive Heart Disease in patients with hypertension. In patients with Hypertensive Heart Disease , abnormalities of both myocardial relaxation and passive filling may be detected sometimes on echocardiography (echo). These diastolic dysfunctions are due to various mechanisms but central to the pathophysiology is an increase in myocardial stiffness. Early symptoms of myocardial stiffness caused by left ventricular hypertrophy (LVH) is a good early indicator for cardiovascular target organ damage in patients with HT and Hypertensive Heart Disease . Hypertensive Heart Disease patients constitute a group in which intensive BP treatment with drugs to strict targets are shown to yield favourable benefit risk ratios. As such, the identification of Hypertensive Heart Disease patients becomes paramount.

An electrocardiogram (ECG) monitors and records the heart's electrical activity. ECG is insensitive to detect diastolic dysfunction with sensitivity from 12% to 50%. An echo takes a picture of the heart using ultrasound. Echo can be used to diagnose diastolic function, however, no one single echo parameter can make the diagnosis. Multiple echo parameters have been proposed including mitral inflow velocity pattern, pulmonary vein flow patterns and tissue Doppler measurements, but imprecise. Existing ultrasound scans cost in the range of US$300-$600 which are reimbursable under Medicaid (the payer). A coronary angiography examines the flow of blood through the heart by inserting a catheter into the heart. It is too invasive and too costly. Therefore, there is appealing need to have a cheaper non-invasive solution that would be able to detect diastolic function. That will have largest impact on patients management and on payers.

A cheap, non-invasive and sensitive solution that permits detection via auscultation of abnormal heart sounds, indicating stiff heart muscle associated with Hypertensive Heart Disease among HT patients is critically needed. Cardiac auscultation (listening to heart sounds) is possible option as heart sounds are associated with myocardial function and dysfunction .In a normal heart, two heart sounds (S1 and S2) are audible, corresponding to closure of the mitral and aortic heart valves respectively. A third heart sound S3, occurring after S2 is present in some heart failure. A fourth heart sound S4, occurring just before S1, is due to forceful contraction of the atrium to overcome a stiff or hypertrophic left ventricle . Human ears are not well equipped to detect such abnormities consistently with a conventional stethoscope. Therefore, investigators propose to develop a low power, non-invasive, portable device which is based on Wireless Sensor Node (WSN) technology to achieve our goal of portable auscultation.Proposed device will allow a monitoring/recording of heart sounds in-situ and perform preliminary assessment of diastolic function that is physiologically meaningful, reproducible and validated. Multiple devices can also be placed and used concurrently at different sites over the torso to enhance chances of detecting abnormal heart sounds.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with clinically suspected or known HT/Hypertensive Heart Disease who have been scheduled for echocardiography examination and/or cardiac catheterization.
2. Participants with history of high BP and stable medication for at least 2 weeks.
3. Presence of the following :

Elevated BP measurement or Left ventricular hypertrophy (LVH) on either prior ECG or prior echo.

Exclusion Criteria for patient

1. Participants with heart muscle disease.
2. Participants with significance valve disease.

Exclusion Criteria for volunteer:

1. Strictly exclude hypertensive for Normal healthy volunteers.
2. Not on any anti-hypertensive agents.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from primary care clinic and outpatient clinics from the National Heart Centre Singapore.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Heart sound measurement from proposed device will be correlated with diastolic functional parameters from echo result and cardiac catheterization. | Through study completion (October 2016)
  Heart sound measurement will be correlated with End diastolic pressure from cardiac catheterisation.

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Tan Ru San, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitworth JA; World Health Organization, International Society of Hypertension Writing Group. 2003 World Health Organization (WHO)/International Society of Hypertension (ISH) statement on management of hypertension. J Hypertens. 2003 Nov;21(11):1983-92. doi: 10.1097/00004872-200311000-00002. PMID 14597836
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Diamond JA, Phillips RA. Hypertensive heart disease. Hypertens Res. 2005 Mar;28(3):191-202. doi: 10.1291/hypres.28.191. PMID 16097361
- [Background] Zannad F, Dousset B, Alla F. Treatment of congestive heart failure: interfering the aldosterone-cardiac extracellular matrix relationship. Hypertension. 2001 Nov;38(5):1227-32. doi: 10.1161/hy1101.099484. PMID 11711528
- [Background] Levy D, Garrison RJ, Savage DD, Kannel WB, Castelli WP. Prognostic implications of echocardiographically determined left ventricular mass in the Framingham Heart Study. N Engl J Med. 1990 May 31;322(22):1561-6. doi: 10.1056/NEJM199005313222203. PMID 2139921
- [Background] Drazner MH, Rame JE, Marino EK, Gottdiener JS, Kitzman DW, Gardin JM, Manolio TA, Dries DL, Siscovick DS. Increased left ventricular mass is a risk factor for the development of a depressed left ventricular ejection fraction within five years: the Cardiovascular Health Study. J Am Coll Cardiol. 2004 Jun 16;43(12):2207-15. doi: 10.1016/j.jacc.2003.11.064. PMID 15193681
- [Background] Lorell BH, Carabello BA. Left ventricular hypertrophy: pathogenesis, detection, and prognosis. Circulation. 2000 Jul 25;102(4):470-9. doi: 10.1161/01.cir.102.4.470. No abstract available. PMID 10908222
- [Background] Marcus GM, Vessey J, Jordan MV, Huddleston M, McKeown B, Gerber IL, Foster E, Chatterjee K, McCulloch CE, Michaels AD. Relationship between accurate auscultation of a clinically useful third heart sound and level of experience. Arch Intern Med. 2006 Mar 27;166(6):617-22. doi: 10.1001/archinte.166.6.617. PMID 16567599
- [Background] Shah SJ, Nakamura K, Marcus GM, Gerber IL, McKeown BH, Jordan MV, Huddleston M, Foster E, Michaels AD. Association of the fourth heart sound with increased left ventricular end-diastolic stiffness. J Card Fail. 2008 Jun;14(5):431-6. doi: 10.1016/j.cardfail.2008.01.010. Epub 2008 May 27. PMID 18514937